CLINICAL TRIAL: NCT06567470
Title: A Phase IIa Double-Blind, Randomized, Parallel-Arm, Placebo-Controlled Trial To Investigate The Effects Of Three Dose Levels Of CIT-013 On Disease Activity In Patients With Moderately Active Rheumatoid Arthritis.
Brief Title: A Study With CIT-013 in RA Patients
Acronym: Citydream
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Citryll BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CITRYLL002
Record Dates: First submitted 2024-08-16; First posted 2024-08-22 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CIT-013 low dose (Experimental): 3 SC injections with low dose CIT-013 and 3 SC injections with medium dose CIT-013
  Interventions: Drug: CIT-013 low dose
- CIT-013 high dose (Experimental): 3 SC injections with CIT-013 high dose and 3 SC injections with CIT-013 medium dose
  Interventions: Drug: CIT-013 high dose
- Placebo (Placebo Comparator): 3 SC injections with placebo and 3 SC injections with CIT-013 medium dose
  Interventions: Drug: Placebo
- CIT-013 medium dose (Experimental): 6 SC injections with CIT-013 medium dose
  Interventions: Drug: CIT-013 medium dose

INTERVENTIONS:
Drug: CIT-013 low dose — Subcutaneous injection
  Arms: CIT-013 low dose
Drug: CIT-013 high dose — Subcutaneous injection
  Arms: CIT-013 high dose
Drug: Placebo — Subcutaneous injection
  Arms: Placebo
Drug: CIT-013 medium dose — CIT-013 medium dose
  Arms: CIT-013 medium dose

SUMMARY:
The goal of this clinical trial is to learn if CIT-013 works to treat rheumatoid arthritis in adults. It will also learn about the safety of CIT-013. The main questions it aims to answer are:

Does CIT-013 lower the disease activity of RA patients? What medical problems do participants have when receiving CIT-013? Researchers will compare CIT-013 to a placebo (a look-alike substance that contains no drug) to see if CIT-013 works to treat the symptoms of RA.

Participants will:

Take receive CIT-013 or placebo every other week for 6 weeks and 50 mg CIT-013 for 6 weeks Visit the clinic once every 2 weeks for checkups and tests Keep monitor their symptoms during this period

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with RA according to the 2010 classification criteria of the American College of Rheumatology (ACR) and the European League Against Rheumatism (EULAR) ≥ 3 months prior to screening
* Aged 18-85
* DAS28-CRP ≥ 3.2, with ≥ 3 Swollen Joints, and ≥ 3 Tender Joints, and CRP ≥ ULN at screening and confirmed prior to randomization
* Stable on a conventional synthetic disease modifying antirheumatic drug for ≥ 4 weeks (csDMARD). This drug must have been used for ≥ 3 months.

Exclusion Criteria:

* High clinical activity or disease severity requiring the immediate start of a biological DMARD (bDMARD) or targeted synthetic DMARD (tsDMARD).
* Contra-indication for CIT-013
* Current inflammatory joint disease other than RA (Sjogren with active disease is included).
* The washout period for bDMARD or JAKi prior to the first dose of investigational product should be at least:

  1. ≥ 1 week for etanercept;
  2. ≥ 4 weeks for adalimumab, infliximab, certolizumab, golimumab, abatacept, tocilizumab, and sarilumab;
  3. ≥ 6 months year for rituximab;
  4. ≥ 2 weeks for tsDMARD (either investigational or commercially available treatment).
* Treated with ≥ 3 bDMARD or tsDMARD
* Injectable corticosteroids or treatment with > 10 mg/day dose of oral prednisolone or equivalent within 4 weeks prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
The change in DAS28-CRP at week 6 compared to baseline | week 6
  Efficacy of CIT-013

SECONDARY OUTCOMES:
Incidence of TEAEs as assessed by CTCAE | 12 weeks
  Safety and tolerability of CIT-013
Maximum Plasma Concentration of CIT-013 before doses | 4, 6, 10 and 12 weeks
  CIT-013 levels

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Kraan, Study Director — Citryll BV
Locations (23):
- Belgium (2):
  - BE-02, Antwerp
  - Site BE-01, Leuven
- Germany (5):
  - DE-04, Bamberg
  - DE-05, Berlin
  - DE-01, München
  - DE-02, München
  - DE-03, Ratingen
- Netherlands (5):
  - NL-02, Amsterdam
  - NL-05, Leeuwarden
  - NL-04, Leiden
  - NL-03, Nijmegen
  - NL-01, Rotterdam
- Poland (5):
  - PL-01, Bialystok
  - PL-03, Lublin
  - PL-02, Poznan
  - PL-05, Torun
  - PL-04, Warsaw
- Spain (6):
  - ES-02, A Coruña
  - ES-04, Barcelona
  - ES-05, Barcelona
  - ES-06, Madrid
  - ES-01, Santander
  - ES-03, Santiago de Compostela